CLINICAL TRIAL: NCT00319033
Title: Long-term Open-label Study in Patients With Interstitial Lung Disease Associated With Systemic Sclerosis Who Completed the Protocol AC-052-330.
Brief Title: Open-label Study With Bosentan in Interstitial Lung Disease
Acronym: BUILD 2 OL
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC-052-332; BUILD 2 OL
Record Dates: First submitted 2006-04-26; First posted 2006-04-27 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Interstitial Lung Disease; Scleroderma
Keywords: interstitial lung disease; scleroderma; bosentan
MeSH Terms: conditions — Lung Diseases, Interstitial; Scleroderma, Diffuse | interventions — Bosentan

INTERVENTIONS:
Drug: bosentan

SUMMARY:
This study will asses the long term safety and efficacy of oral bosentan to patients suffering from Interstitial Lung Disease.

ELIGIBILITY:
Inclusion Criteria:

* To have completed the 12-month treatment period of the AC-052-330/BUILD 2.
* Women should not be pregnant
* Women of childbearing potential must have a negative pre-treatment pregnancy test and use a reliable method of contraception
* Signed informed consent prior to initiation of any study-mandated procedure

Exclusion Criteria:

* Any major violation of the protocol AC-052-330.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 132
Dates: Start 2004-07; Primary Completion 2006-02 (Actual); Study Completion 2006-02 (Actual)

PRIMARY OUTCOMES:
Change from baseline to all assessed time points in 6-minute walk test distance.
Change from baseline to all assessed time points in Borg dyspnea index, FVC and DLco, SpO2 at rest and de-saturation index (6-minute walk distance multiplied by SpO2 mean value).
Transition Dyspnea Index at all assessed time points.
Change from baseline to all assessed time points in SpO2 mean value, time to de-saturation (decrease in SpO2 ≥ 4%), trough SpO2 and area under the curve during 6-minute walk test.

SECONDARY OUTCOMES:
Adverse events; serious adverse events.